CLINICAL TRIAL: NCT06916793
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel-group Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-843 in Male Patients With Androgenetic Alopecia
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy of CKD-843 in Male Patients With Androgenetic Alopecia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A107_03AGA2318
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group1 (Experimental): CKD-843 dose#1 + Placebo of Dutasteride Capsule
  Interventions: Drug: CKD-843 dose#1; Drug: Placebo of Dutasteride Capsule
- Test Group2 (Experimental): CKD-843 dose#2 + Placebo of Dutasteride Capsule
  Interventions: Drug: CKD-843 dose#2; Drug: Placebo of Dutasteride Capsule
- Placebo-controlled Group (Placebo Comparator): Placebo of CKD-843 dose + Placebo of Dutasteride Capsule
  Interventions: Drug: Placebo of CKD-843 dose; Drug: Placebo of Dutasteride Capsule
- Active-controlled Group (Active Comparator): Placebo of CKD-843 dose + Dutasteride Capsules
  Interventions: Drug: Placebo of CKD-843 dose; Drug: Dutasteride Capsules

INTERVENTIONS:
Drug: CKD-843 dose#1 — IM injection every 3 months for 12 months
  Arms: Test Group1
Drug: CKD-843 dose#2 — IM injection every 3 months for 12 months
  Arms: Test Group2
Drug: Placebo of CKD-843 dose — IM injection every 3 months for 12 months
  Arms: Active-controlled Group; Placebo-controlled Group
Drug: Dutasteride Capsules — oral, once daily, 12 months
  Arms: Active-controlled Group
Drug: Placebo of Dutasteride Capsule — oral, once daily, 12 months
  Arms: Placebo-controlled Group; Test Group1; Test Group2

SUMMARY:
This is a multi-centers, randomized, double-blind, parallel-group, Phase 3 Trial to evaluate the efficacy and safety of CKD-843 in Male patients with Androgenetic Alopecia

DETAILED DESCRIPTION:
The participants were randomly assigned to one of the following groups: CKD-843 dose #1, CKD-843 dose #2, placebo, or Dutasteride group. They received the assigned medication, placebo for blinding, or the reference drug over a 12-month period.

ELIGIBILITY:
Key Inclusion Criteria:

* Male of age 18-50 years
* Clinical Diagnosis of Androgenetic Alopecia
* Written informed consent

Key Exclusion Criteria:

* Other types of Alopecia or other diseases that can cause hair loss
* Clinically significant scalp disease such as seborrheic dermatitis or psoriasis
* Clinically significant hepatic disease, thyroid disease, or mental illness, as determined by the Investigator
* Participants who do not agree to use contraception during the trial and for 24 weeks after the last dose, and plan to provide sperm or conceive within 24 weeks after the last dose

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-12-19 (Estimated); Study Completion 2027-09-17 (Estimated)

PRIMARY OUTCOMES:
Total number of hair Changes | Baseline, Week 24
  from Baseline at Week24 of total number of hair changes

CONTACTS AND LOCATIONS:
Overall Officials: OhSang Kwon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No